CLINICAL TRIAL: NCT04437121
Title: Dietary and Lifestyle Habits of Children and Adolescents and Their Parents During the Pandemic of COVID-19 in Greece: The COV-EAT Study
Brief Title: Dietary and Lifestyle Habits During the Pandemic of COVID-19 in Greece
Acronym: COV-EAT
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Odysseas Androutsos, Odysseas Androutsos, M.Med.Sci., Ph.D. Associate Professor, Department of Nutrition-Dietetics, Univ. of Thessaly, University of Thessaly
Other Study IDs: COV-EAT
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Eating Behavior; COVID-19
Keywords: Eating Habits; Sedentary Behavior; Childhood Obesity; Quarantine; COVID-19; School Closings
MeSH Terms: conditions — Feeding Behavior; COVID-19; Sedentary Behavior; Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents of children aged 2-18 years: Parents of children aged 2-18 years during the lockdown due to the COVID-19 pandemic, following their informed consent form prior to their participation to the study.
  Interventions: Other: Online Survey about Dietary and Lifestyle Habits

INTERVENTIONS:
Other: Online Survey about Dietary and Lifestyle Habits — An online survey was conducted in a random sample of families. Parents self-reported their child's and their own dietary and lifestyle habits, as well as information about their sociodemographic status.
  The survey consisted of 70 questions in 3 sections.

SUMMARY:
The aim of this study was to examine potential changes in children' and adolescents' dietary and lifestyle (physical activity, sedentary behaviour and sleep) habits during the quarantine that was implemented in Greece due to COVID-19. An online survey in a random sample of families across Greece was conducted. Parents self-reported their children's and their own dietary and lifestyle habits, as well as information about their sociodemographic status.

DETAILED DESCRIPTION:
Since December 2019, the world is facing a new disease (COVID-19), which is caused by the Coronavirus (Sars CoV-2). WHO declared the disease of COVID-19 as a pandemic in February 2020. Since then, many countries around the world have imposed lockdown (quarantine at home), as the main measure to prevent the spreading of the disease. In Greece, the lockdown was officially imposed from March, 23rd, 2020. This unprecedented situation may have caused changes in adults' and children's dietary and lifestyle habits.

Data were collected via an online survey consisting of 70 questions. Study participants were enrolled after signing an informed consent form. The questionnaire self-reported by volunteers (parents of children aged between 2-18 years old). The survey had 3 sections. The first section focused on participants' sociodemographic data (e.g. gender, age, city of residence and socioeconomic level). The second and third sections contained questions about the parents' (section 2) and their children's (section 3) dietary and lifestyle habits before and during quarantine.

The scientific community raises concerns about the health implications that will be caused due to the COVID-19 lockdown. The results of this study are expected to shed light into children and adolescents, as well as their parents', changes in dietary and lifestyle behaviours and feed the development of effective strategies to prevent the adoption of unhealthy lifestyle behaviours and weight gain in the event of a second wave of COVID-19 in the coming months.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of children and adolescents, aged 2-18 years.
2. During the lockdown period due to the COVID-19 pandemic in Greece.
3. Parents signed an informed consent form prior to their participation to the study

Exclusion Criteria:

1. Parents of children <24 months old.
2. Parents of children >18 years old.
3. Parents not living in Greece.
4. Parents who did not sign the consent form.

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Parents of children and adolescents, aged 2-18 years, during the lockdown period due to the COVID-19 pandemic in Greece.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-05-24 (Actual); Study Completion 2020-05-24 (Actual)

PRIMARY OUTCOMES:
Change in weight (child) | Approximately one month before the Greek lockdown period (February 2020) and two months during the quarantine period (23 March 2020 till 24 May 2020)
  Weight in kg will be measured using scales at home
Behaviour (child) | Approximately one month before the Greek lockdown period (February 2020) and two months during the quarantine period (23 March 2020 till 24 May 2020)
  Eating Behaviour during the quarantine, measured with an online (FFQ) questionnaire.

SECONDARY OUTCOMES:
Behaviour (parents) | Approximately one month before the Greek lockdown period (February 2020) and two months during the quarantine period (23 March 2020 till 24 May 2020)
  Eating Behaviour during the quarantine, measured with an online questionnaire.
Physical Activity Levels (child) | Approximately two months before the Greek lockdown period (January-February 2020) and two months during the quarantine period (23 March 2020 till 24 May 2020)
  Child's physical activity levels during the quarantine period, measured with an online questionnaire.
Screen Time (child) | Approximately two months before the Greek lockdown period (January-February 2020) and two months during the quarantine period (23 March 2020 till 24 May 2020)
  Changes in children' screen time (hours per day) during the quarantine period, measured with an online questionnaire.
Sleep Duration (child) | Approximately two months before the Greek lockdown period (January-February 2020) and two months during the quarantine period (23 March 2020 till 24 May 2020)
  Changes in children' sleep time (hours per day) during the quarantine period, measured with an online questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Odysseas Androutsos, M.Med.Sci., Ph.D., Principal Investigator — University of Thessaly
Locations (1):
- Department of Nutrition-Dietetics, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided
All IPD that underlie results in a publication

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04437121/Prot_SAP_ICF_000.pdf